CLINICAL TRIAL: NCT01654627
Title: Horizontal Guided Bone Regeneration for Dental Implants Using Synthetic Membrane (Regenecures' AMCA GBR Dental Membrane) a Prospective, Randomized,Controlled Study.
Brief Title: Guided Bone Regeneration Using Synthetic Membrane
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RegeneCure, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGD001
Record Dates: First submitted 2012-07-26; First posted 2012-08-01 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Jaw, Edentulous; Jaw, Edentulous, Partially
Keywords: Guided Tissue Regeneration; Dental Implants; Membrane, Synthetic
MeSH Terms: conditions — Jaw, Edentulous; Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regenecure AMCA GBR Dental membrane (Experimental): 16 patients will undergo the guided bone regeneration procedure using the Regenecure AMCA Membrane
  Interventions: Device: Regenecure AMCA GBR Dental Membrane
- Collagen membrane (Active Comparator): 16 patients will undergo the guided bone regeneration procedure using a commercially available collagen membrane
  Interventions: Device: Geistlich Bio-Gide® collagen membrane

INTERVENTIONS:
Device: Regenecure AMCA GBR Dental Membrane — Patients will undergo Guided Bone Regeneration (GBR) procedure using the Regenecure AMCA GBR Membrane
  Arms: Regenecure AMCA GBR Dental membrane
Device: Geistlich Bio-Gide® collagen membrane — The Geistlich Bio-Gide® collagen membrane, a commercially available product, will be used in 10 patients.
  Arms: Collagen membrane

SUMMARY:
The purpose of this study is to examine the safety and usefulness of the Regenecure guided bone regeneration membrane for stimulating bone growth in patients that don't have enough bone for dental implant placement. The study will include 16 patients in each group, 20 non-smokers and 12 smokers, a total of 32 patients will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have voluntarily signed the informed consent form before any study related action
* Age: 18 to 65 with missing teeth, seeking for implant therapy.
* Men/Women
* In good systemic health
* Present with no contra indication against oral surgical interventions
* Single/ multiple tooth gap - have at least one missing tooth in the mandible or maxilla, requiring one or more dental implants.
* The tooth at the implant site(s) must have been extracted or lost at least 6 weeks before the date of implantation.
* Bone defect(s) must be present with a lateral dimension greater than or equal to 5 mm or less.
* Full mouth plaque score (FMPI) lower or equal than 25%
* Patients must be committed to the study

Exclusion Criteria:

* Medical conditions requiring prolonged use of steroids
* Use of Bisphosphonate intravenously
* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Immunocompromised patients
* Uncontrolled Diabetes
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.
* Untreated inflammation
* Mucosal diseases or oral lesions
* History of local irradiation therapy
* Persistent intraoral infection
* Patients with bad oral hygiene or unmotivated for normal home care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Bone volume | Change from Baseline in bone volume at 6 months
  Clinical effect on bone volume measured using CBCT. The volume of the newly formed bone will be evaluated by "subtraction" of the 2 cone beam CTs using digital measurements.

SECONDARY OUTCOMES:
Histomorphometry | 6 months
  Specimens will be prepared for histological staining (H&E and Masson's trichrome stain). The stained samples will be evaluated for new bone, residual bone graft, marrow spaces and vascularity.
Safety will be demonstrated by using VAS scale for pain measurements and if the PI will consider that any adverse event device related isn't clinically significant | six months
  Safety will be demonstrated by using VAS scale for pain measurements and if the PI will consider that any adverse event device related isn't clinically significant

CONTACTS AND LOCATIONS:
Overall Officials: Lior Shapira, PhD, Principal Investigator — Haddasah Medical Center, Jerusalem Israel
Locations (1):
- Department of Periodontology Hadassah and Hebrew University Medical Center, Jerusalem, Israel